CLINICAL TRIAL: NCT03921151
Title: 5-HT2AR: 5HT2CR Balance in Brain Connectivity in Cocaine Dependence
Brief Title: 5HT2CR Balance in Brain Connectivity in Cocaine Dependence
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: The University of Texas Medical Branch, Galveston (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: HM15289; P20DA024157-04S1 (NIH)
Record Dates: First submitted 2019-04-10; First posted 2019-04-19 (Actual); Results first posted 2021-11-22 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Cocaine Dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Mirtazapine; Tablets

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cocaine-dependent (Other): Participants who use and are dependent on cocaine
  Interventions: Drug: Mirtazapine 15 MG Oral Tablet
- Non-drug using Healthy Controls (Other): Participants who are not drug users
  Interventions: Drug: Mirtazapine 15 MG Oral Tablet

INTERVENTIONS:
Drug: Mirtazapine 15 MG Oral Tablet — The intervention will be a 15mg of mirtazapine oral tablet given to participants prior to their treatment scan and assessments. In order to ensure that biases or social desirability do not contaminate baseline assessments, all participants will also be given a tablet consisting of dextrose in gelatin prior to their baseline scan and assessment.
  Other Names: Remeron

SUMMARY:
This project will evaluate the role of the 5-HT2CR:5-HT2AR balance in impulsive action and cue reactivity in cocaine-dependent subjects as compared to non-drug using controls.

DETAILED DESCRIPTION:
The overall goal of this project is to evaluate the role of molecular interactions between 5-HT2AR and 5-HT2CR in behavioral phenotypes that confer risk for cocaine dependence and relapse. Specifically, this project will evaluate the role of the 5-HT2CR:5-HT2AR balance in impulsive action and cue reactivity in cocaine-dependent subjects as compared to non-drug using controls. Brain and behavioral responses to the 5-HT2AR blocking medication mirtazapine will be compared between subjects who have high and low functioning of the 5-HT2CR based on presence of a specific, functionally-relevant single nucleotide polymorphism (SNP) of the 5-HT2CR (Cys23Ser). The 5-HT2CR Cys23Ser SNP is thought to decrease the function of the protein and a preliminary observation indicates cocaine-dependent subjects carrying the CC genotype (Ser23 protein variant) display significantly higher cue reactivity. For Aims 1 and 2, two fMRI analysis methods will be used: 1) a voxelwise whole brain analysis; 2) a region of interest analysis based on proposed integrative circuitry shown in the model below. Because neuroimaging studies have shown that performance of impulsive action tasks and exposure to cocaine-associated cues (cue reactivity paradigms) activate brain regions in brain circuits in humans, impulsive action and cue reactivity may be engendered in related pathways. To explore this hypothesis, researchers will employ functional magnetic resonance imaging (fMRI)-based dynamic causal modeling (DCM) to ascertain the causal influences of one brain region over another. Employing DCM, researchers will uncover the effective connectivity within nodes of the neurocircuitry involved in impulsive action and cue reactivity. This project will parallel preclinical work studying the relationship between 5-HT2AR and 5-HT2CR on impulsive action and cue reactivity.

ELIGIBILITY:
Inclusion Criteria:

Cocaine Dependent Subjects

1. Be English-speaking volunteers
2. Be aged between 18 and 60 years
3. Meet DSM-5 criteria for cocaine dependence
4. Have a self-reported history of using cocaine
5. Have hematology and chemistry laboratory tests that are within reference limits ( 10%) with the following exceptions: hemoglobin and hematocrit within normal limits (for fMRI).
6. Have a baseline EKG that demonstrates clinically normal sinus rhythm, clinically normal conduction, and no clinically significant abnormalities
7. Have a medical history and physical examination demonstrating no clinically significant contraindications for study participation, in the judgment of the admitting physician and the principal investigator.
8. Have no metal fragments or other bodily metal (e.g., pacemaker) or significant claustrophobia that would put the subjects at risk for MRI scanning.

Non-Drug Using Controls

1. Be English-speaking volunteers
2. Be aged between 18 and 60 years
3. Have no past history of Psychiatric or non-Psychiatric medical disorders which could affect the central nervous system as assessed by SCID and physical examination.
4. Have hematology and chemistry laboratory tests that are within reference limits ( 10%), with the following exceptions: hemoglobin and hematocrit within normal limits (for fMRI)
5. Have a baseline EKG that demonstrates clinically normal sinus rhythm, clinically normal conduction, and no clinically significant abnormalities
6. Have a medical history and brief physical examination demonstrating no clinically significant contraindications for study participation, in the judgment of the admitting physician and the Principal investigator.
7. Have no metal fragments or other bodily metal (pacemaker) or significant claustrophobia that would put the subjects at risk for MRI scanning

Exclusion Criteria:

Cocaine Dependent Subjects

1. Have any history or evidence suggestive of seizure disorder or brain injury.
2. Have any previous medically adverse reaction to mirtazapine or other antidepressants.
3. Have neurological or psychiatric disorders, such as (a) psychosis, bipolar illness or major depression as assessed by SCID; (b) organic brain disease or dementia assessed by clinical interview; (c) history of any psychiatric disorder that would require ongoing treatment or that would make study compliance difficult; and (d) history of suicide attempts within the past 3 months and/or current suicidal ideation/plan.
4. Have evidence of uncontrolled clinically significant heart disease or hypertension, as determined by the PI.
5. Have evidence of non-psychiatric medical illness including neuroendocrine, autoimmune, renal, hepatic, or active infectious disease.
6. Use of any medications or drugs that can affect the central nervous system other than cocaine, marijuana, alcohol caffeine and nicotine.
7. Have a positive HIV test.
8. Be pregnant or nursing. Other females must either be unable to conceive (i.e., surgically sterilized, sterile, or postmenopausal) or be using a reliable form of contraception (e.g., abstinence, birth control pills, intrauterine device, condoms, or spermicide). All females must provide negative pregnancy urine tests before study entry, weekly during the study, and at the end of study participation.
9. Have any other illness, condition, or use of psychotropic medications, which in the opinion of the PI and/or the admitting physician would preclude safe and/or successful completion of the study.

Non-Drug Using Controls

1. Meet DSM-5 criteria for any current or past Axis I disorder.
2. Meet DSM-5 criteria for an Axis II diagnosis of Borderline or Antisocial Personality Disorder.
3. Have any history or evidence suggestive of seizure disorder or brain injury.
4. Have any previous medically adverse reaction to mirtazapine or other antidepressants.
5. Have evidence of uncontrolled clinically significant heart disease or hypertension, as determined by the PI.
6. Have evidence of medical illness including neuroendocrine, autoimmune, renal, hepatic, or active infectious disease.
7. Use of any medications or drugs that can affect the central nervous system other than caffeine or nicotine.
8. Have a positive HIV test.
9. Be pregnant or nursing. Other females must either be unable to conceive (i.e., surgically sterilized, sterile, or postmenopausal) or be using a reliable form of contraception (e.g., abstinence, birth control pills, intrauterine device, condoms, or spermicide). All females must provide negative pregnancy urine tests before study entry, weekly during the study, and at the end of study participation.
10. Have any other illness, condition, or use of psychotropic medications, which in the opinion of the PI and/or the admitting physician would preclude safe and/or successful completion of the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2014-05-13 (Actual); Primary Completion 2019-01-24 (Actual); Study Completion 2019-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Moeller, M.D., Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cocaine-dependent | Non-drug Using Healthy Controls
Started | 46 | 44
Completed | 35 | 28
Not Completed | 11 | 16
Not completed — Withdrawal by Subject | 11 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cocaine-dependent | Non-drug Using Healthy Controls | Total
Number analyzed (Participants) | 35 | 28 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.6 (8.62) | 34.29 (12.5) | 40.02 (11.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 14 | 23
  Male | 26 | 14 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 35 | 28 | 63
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 34 | 24 | 58
  White | 1 | 4 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 35 | 28 | 63

OUTCOME MEASURES:

1. Primary Outcome: Change in Interaction of the Serotonin Receptor (5-HTR) Type-2C Cys23Ser Single Nucleotide Polymorphism (SNP) and a 5-HT2AR Antagonist on the Functional Circuitry Underlying Impulsive Action.
Description: Change in fMRI activation during Go/NoGo (impulsivity) task with placebo dose vs Mirtazapine dose.
  Brain activation measured using blood-oxygen-level dependent (BOLD) contrast
Time Frame: Baseline to 1 week
Population: Change scores could not be calculated for 17 cocaine-dependent participants and 14 non-drug using participants due to a missing or unusable fMRI scan.
Measure: Mean (90% Confidence Interval); unit: percent of whole brain BOLD signal
Arm/Group | Cocaine-dependent | Non-drug Using Healthy Controls
Number analyzed (Participants) | 18 | 14
percent of whole brain BOLD signal | 0.6889 [0.2164 to 1.1614] | -1.1091 [-1.9063 to -0.3119]

2. Secondary Outcome: Change in Interaction of the 5-HT2CR Cys23Ser SNP and a 5-HT2AR Antagonist on the Functional Circuitry Underlying Cue Reactivity
Description: Change in fMRI activation during Attentional bias task with placebo dose vs Mirtazapine dose measured using whole brain blood oxygenation level dependent (BOLD) signal
Time Frame: Baseline to 1 week
Population: Change scores could not be calculated for 12 cocaine-dependent participants and 9 non-drug using participants due to a missing or unusable fMRI scan.
Measure: Mean (90% Confidence Interval); unit: percent of BOLD signal
Arm/Group | Cocaine-dependent | Non-drug Using Healthy Controls
Number analyzed (Participants) | 23 | 19
percent of BOLD signal | -0.135 [-0.2998 to 0.0298] | 0.2225 [-0.0926 to 0.5377]

3. Other Pre Specified Outcome: Change in Effective Connectivity Involved in the 5-HT2AR:5-HT2CR Homeostasis Impulsive Action
Description: Change in Impulsivity as measured by Go/NoGo task with placebo dose vs Mirtazapine dose
Time Frame: Baseline to 1 week
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Change in Effective Connectivity Involved in the 5-HT2AR:5-HT2CR Homeostasis Cue Reactivity
Description: Change in Cue reactivity as measured by Attentional bias task with placebo dose vs Mirtazapine dose
Time Frame: Baseline to 1 week
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Change in Explore Interactions Between Other 5-HT2CR SNPs and Brain Activation During Attentional Bias Task After a 5- HT2AR Antagonist
Description: Change in fMRI activation with other 5-HT2CR SNPs during Attentional bias task with placebo dose vs Mirtazapine dose
Time Frame: Baseline to 1 week
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Change in Explore Interactions Between Other 5-HT2CR SNPs and Brain Activation During Go/NoGo (Impulsivity) Task After a 5- HT2AR Antagonist
Description: Change in fMRI activation with other 5-HT2CR SNPs during Go/NoGo (impulsivity) task with placebo dose vs Mirtazapine dose
Time Frame: Baseline to 1 week
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were monitored during the first study visit (practice MRI) through the last study visit (Dose 2 MRI) approximately 1 week.
Description: During the practice MRI visit, adverse events (AEs) were recorded using the 24 hour questionnaire. During the Dose 1 and Dose 2 MRI visits, AEs were recorded using the 24 questionnaire (pre dose), Drug Effects Questionnaire (pre dose, 1.25 hr post dose, 3.75 hr post dose, 4.5 hr post dose), and neurological exam (5 hr post dose completed by physician). All AEs were entered into a secure REDCap database.
Arm/Group | Cocaine-dependent | Non-drug Using Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/28
Other Adverse Events (participants affected / at risk) | 0/35 | 1/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cocaine-dependent (N=35) | Non-drug Using Healthy Controls (N=28)
Nausea and dizziness (Gastrointestinal disorders) | 0 (0) | 1 (1) — During mirtazapine administration

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-11): https://cdn.clinicaltrials.gov/large-docs/51/NCT03921151/Prot_SAP_001.pdf
  • Informed Consent Form (2019-09-11): https://cdn.clinicaltrials.gov/large-docs/51/NCT03921151/ICF_002.pdf